CLINICAL TRIAL: NCT04079140
Title: Benefits of Self-administered Vaginal Dinoprostone Administration 12 Hours Prior to Intrauterine Device Insertion in Adolescent and Young Women: a Randomized Controlled Trial
Brief Title: Vaginal Dinoprostone Administration Prior to Intrauterine Device Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vaginal dinoprostone IUD
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: IUD Insertion Pain
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) self-inserted by the patient 12 hours before IUD insertion.
  Interventions: Drug: Dinoprostone
- placebo (Placebo Comparator): one tablet of placebo self-administered by the patient 12 hours before IUD insertion.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) self-inserted by the patient 12 hours before IUD insertion.
  Arms: dinoprostone
Drug: placebo — one tablet of placebo self-inserted by the patient 12 hours before IUD insertion.
  Arms: placebo

SUMMARY:
To investigate whether vaginal dinoprostone administered before the levonorgestrel-releasing intrauterine system(IUs) insertion reduces IUD insertion pain and difficulty in insertion in adolescents and young women.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous adolescent and young women requesting levonorgestrel-releasing intrauterine device

Exclusion Criteria:

* pregnancy and contraindication or allergy to dinoprostone or contraindication to IUD insertion, chronic pelvic pain,pelvic inflammatory disease,analgesic intake 24 hours prior to IUD insertion.

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Giza, Egypt